CLINICAL TRIAL: NCT02507349
Title: Amplifying the Patient's Voice: Person-Centered Versus Measurement-Based Approaches in Mental Health
Brief Title: Person-Centered Versus Measurement-Based Care in Mental Health
Acronym: PCORI-SDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Dartmouth College (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Kim MacDonald-Wilson, Senior Director, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CDR-1306-02474
Record Dates: First submitted 2015-06-30; First posted 2015-07-23 (Estimated); Results first posted 2019-02-01 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Schizophrenia; Bipolar Disorder; Major Depression
Keywords: serious mental illness; mental health services research; measurement-based care; shared decision making; psychiatric medication management; community psychiatry; comparative effectiveness research; mixed methods research
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Depressive Disorder, Major | interventions — Patient-Centered Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Person-Centered Care (Active Comparator): Decision support center staffed by peers. Patient uses the CommonGround program prior to medication visit to prepare a personal report, with support from peer(s). The CommonGround report expresses goals for medication, how other strategies help with functioning, current problems, and medication side effects. Patient brings report into the medication visit. Prescriber and patient discuss medication options, and prescriber enters the shared decision into CommonGround during the visit.
  Interventions: Behavioral: Person-Centered Care
- Measurement-Based Care (Active Comparator): Clinic staff asks each patient to use a tablet computer to complete a brief assessment of symptoms and problems prior to medication visit. Prescriber views assessment results on office computer and discusses next steps in medication management with the patient.
  Interventions: Behavioral: Measurement-Based Care

INTERVENTIONS:
Behavioral: Person-Centered Care — Decision support center staffed by peers. Patient uses the CommonGround program prior to medication visit to prepare a personal report, with support from peer(s). The CommonGround report expresses goals for medication, how other strategies help with functioning, current problems, and medication side effects. Patient brings report into the medication visit. Prescriber and patient discuss medication options, and prescriber enters the shared decision into CommonGround during the visit.
  Arms: Person-Centered Care
Behavioral: Measurement-Based Care — Clinic staff asks each patient to use a tablet computer to complete a brief assessment of symptoms and problems prior to medication visit. Prescriber views assessment results on office computer and discusses next steps in medication management with the patient.
  Arms: Measurement-Based Care

SUMMARY:
Fifteen minutes is the typical length of an outpatient medication management appointment for people with serious mental health conditions. These brief interactions with prescribers are frequently provider-driven with insufficient time focused on the patient's needs and personal recovery. Shared decision making is a strategy that could improve this interaction. This study examines how technology can be used in the care process to amplify the voice of the patient, support shared decisions, and improve treatment outcomes.

Investigators will compare the effectiveness of Measurement-Based vs. Person-Centered Care on two primary patient-centered outcomes: the patient experience of care with medication treatment and the level of shared decision making. Investigators hypothesize that:

1. Person-Centered Care will result in greater improvement in patient experience of care with medication treatment than Measurement-Based Care.
2. Person-Centered Care will result in a greater level of shared decision making during the medication visit than Measurement-Based Care.

The study team will collect information from patients, caregivers, and clinic staff at different points in time during the study. Patients will be asked to complete questionnaires, and additional data on their service use will be gathered. Some patients and providers will also be interviewed about their experiences with care. Investigators are especially interested to learn if and how these two approaches are perceived to change medication treatment, if patients are more satisfied and empowered in their care, and why and how providers perceive and adopt changes to their clinical care.

DETAILED DESCRIPTION:
An important attribute of patient-centered care is the active engagement of patients in making health care decisions. Despite advances in health care to support shared decision making, the patient experience of mental health care remains provider-driven. For individuals with serious mental illness (SMI), important decisions involve the choice of medications and how best to use medications to support individualized, person-centered recovery goals. By comparing the effectiveness of two approaches for promoting shared decision making around medication treatment on outcomes that matter most to individuals with SMI, the proposed study will advance ongoing and much-needed efforts to evolve toward a more personalized, recovery-oriented system of mental health care.

Building on the work of a multi-stakeholder collaboration, investigators will compare two interventions, Person-Centered Care and Measurement-Based Care, both focused on patient-prescriber interactions around medication treatment. The investigators' study will address three questions that patients have identified as important to them:

1. Are there ways I can be more involved in my care that will result in better outcomes?
2. How likely am I to benefit from improved communication with my prescriber?
3. How will shared decision making support my personal recovery and overall wellness?

Study aims will compare the effectiveness of measurement-based vs. person-centered care on the patient experience of care and on shared decision making. Investigators hypothesize that:

1. Person-Centered Care will result in greater improvement in patient experience of care with medication treatment than Measurement-Based Care.
2. Person-Centered Care will result in a greater level of shared decision making during the medication visit than Measurement-Based Care.

In addition, investigators will compare the effectiveness of the two approaches on seven secondary patient-centered outcomes, and examine differences in outcomes within the two approaches for subgroups of patients based on their: (1) current status regarding psychiatric medication, (2) engagement with the interventions, and (3) illness severity.

The target population is 2,460+ Medicaid-enrolled adults with SMI who receive medication treatment at one of 15 community mental health centers (CMHC). Using a prospective cluster-randomized design with a mixed-methods approach, investigators will randomly assign CMHCs to one of the two interventions. Quantitative (self-report, claims, process) and qualitative (interviews) data will be gathered at multiple time points across the two-year intervention period (baseline, 8 months, 16 months, and 24 months). Multi-level longitudinal analyses will examine the impact of the interventions on outcomes and explore the role of moderating variables. Qualitative data will be used to understand patient and stakeholder perspectives and to promote dissemination and sustainability.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 and older
* Non-SMI (anxiety, post-traumatic stress disorder, depression, dysthymia, depression NOS) or SMI (schizophrenia, bipolar disorder, major depression)
* Receiving services at one of the 15 participating community mental health centers
* At least three claims for medication management services in past 12 months
* Insured by Community Care Behavioral Health Organization

Exclusion Criteria:

* Assessed by clinicians as being too ill to be treated on an outpatient basis
* Unable to speak, read, or understand English at the minimum required level

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2443 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2017-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory J McHugo, PhD, Principal Investigator — Dartmouth Psychiatric Research Center, The Geisel School of Medicine at Dartmouth; Kim MacDonald-Wilson, ScD,CRC,CPRP, Principal Investigator — UPMC Center for High-Value Health Care; Patricia E Deegan, PhD, Principal Investigator — Pat Deegan, PhD & Associates, LLC
Locations (2):
- United States (2):
  - Dartmouth Psychiatric Research Center, Lebanon, New Hampshire
  - UPMC Center for High-Value Health Care, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Person-Centered Care: Decision support center staffed by peers. Patient uses the CommonGround program prior to medication visit to prepare a personal report, with support from peer(s). The CommonGround report expresses goals for medication, how other strategies help with functioning, current problems, and medication side effects. Patient brings report into the medication visit. Prescriber and patient discuss medication options, and prescriber enters the shared decision into CommonGround during the visit.
  Person-Centered Care: Decision support center staffed by peers. Patient uses the CommonGround program prior to medication visit to prepare a personal report, with support from peer(s). The CommonGround report expresses goals for medication, how other strategies help with functioning, current problems, and medication side effects. Patient brings report into the medication visit. Prescriber and patient discuss medication options, and prescriber enters the shared decision into CommonGround during the visi
Period: Overall Study
Arm/Group | Person-Centered Care | Measurement-Based Care
Started | 1232 | 1211
Completed | 1045 | 1050
Not Completed | 187 | 161
Not completed — Death | 12 | 16
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 174 | 144

BASELINE CHARACTERISTICS:
Population: The analysis population is different from the assignment in the Participant Flow because participants were only included in analysis if they had a baseline survey record (i.e., not all who consented completed baseline questionnaires).
Groups:
- Total: Total of all reporting groups
Arm/Group | Person-Centered Care | Measurement-Based Care | Total
Number analyzed (Participants) | 1201 | 1162 | 2363
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.82 (12.41) | 41.31 (11.88) | 41.57 (12.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 716 | 775 | 1491
  Male | 485 | 387 | 872
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 37 | 14 | 51
  Not Hispanic or Latino | 1164 | 1148 | 2312
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 6 | 2 | 8
  Black/African American | 103 | 104 | 207
  Native American | 7 | 2 | 9
  White | 1015 | 1023 | 2038
  Other | 70 | 31 | 101
Region of Enrollment [Number; unit: participants]
  United States | 1201 | 1162 | 2363

OUTCOME MEASURES:

1. Primary Outcome: Patient Experience of Medication Treatment (PEMM)
Description: The PEMM is a 12-item self-report measure of mental health patient experience of medication management with prescribers .Response options for 11 questions range from 0=Never to 4=Always, and the response options for the final question range from 0=Very Dissatisfied to 4=Very Satisfied. Overall possible range was 0 to 4. PEMM scores for each time point reflect the mean score of all measures collected within that time frame.
Time Frame: Baseline and every eight months during the two-year intervention phase
Population: Multiple records can be measured from the same participant at the same time period, so overall number of surveys analyzed can be greater than the unique number of participants except for at baseline.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: Survey Records
Arm/Group | Person-Centered Care | Measurement-Based Care
Number analyzed (Participants) | 1201 | 1162
Number analyzed (Survey Records) | 3795 | 3772
Units on a scale
  Baseline: number analyzed (Participants) | 1201 | 1161
  Baseline: number analyzed (Survey Records) | 1201 | 1161
  Baseline | 3.009 (0.712) | 3.007 (0.747)
  Month 3: Every record 0< month <=3: number analyzed (Participants) | 5 | 3
  Month 3: Every record 0< month <=3: number analyzed (Survey Records) | 5 | 3
  Month 3: Every record 0< month <=3 | 2.6 (0.91) | 3.09 (0.18)
  Month 6: Every record 3< month <=6: number analyzed (Participants) | 229 | 192
  Month 6: Every record 3< month <=6: number analyzed (Survey Records) | 229 | 192
  Month 6: Every record 3< month <=6 | 3.056 (0.679) | 3.068 (0.675)
  Month 8: Every record 6< month <=8: number analyzed (Participants) | 308 | 246
  Month 8: Every record 6< month <=8: number analyzed (Survey Records) | 308 | 246
  Month 8: Every record 6< month <=8 | 3.015 (0.713) | 3.083 (0.735)
  Month 12: Every record 8< month <=12: number analyzed (Participants) | 268 | 297
  Month 12: Every record 8< month <=12: number analyzed (Survey Records) | 288 | 315
  Month 12: Every record 8< month <=12 | 3.055 (0.715) | 3.119 (0.682)
  Month16: Every record 12< month <=16: number analyzed (Participants) | 541 | 448
  Month16: Every record 12< month <=16: number analyzed (Survey Records) | 766 | 525
  Month16: Every record 12< month <=16 | 3.066 (0.685) | 3.112 (0.681)
  Month 18: Every record 16< month <=18: number analyzed (Participants) | 195 | 366
  Month 18: Every record 16< month <=18: number analyzed (Survey Records) | 204 | 406
  Month 18: Every record 16< month <=18 | 3.134 (0.703) | 3.153 (0.624)
  Month 20: Every record 18< month <=20: number analyzed (Participants) | 331 | 352
  Month 20: Every record 18< month <=20: number analyzed (Survey Records) | 384 | 382
  Month 20: Every record 18< month <=20 | 3.062 (0.666) | 3.113 (0.677)
  Month 24: Every record 20< month: number analyzed (Participants) | 341 | 417
  Month 24: Every record 20< month: number analyzed (Survey Records) | 410 | 492
  Month 24: Every record 20< month | 3.13 (0.667) | 3.117 (0.7)
Statistical Analysis 1: Comparison: Person-Centered Care vs Measurement-Based Care; Time-by-treatment interaction; Test type: Superiority; p < 0.0001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Person-Centered Care vs Measurement-Based Care; Three-way interaction effect (treatment, polynomial time, and age group 1) where age group 1 is defined by 0 (reference) if <=35; 1 if (35<age<=49); 2 if age >49; Test type: Superiority; p = 0.0033, Mixed Models Analysis
Statistical Analysis 3: Comparison: Person-Centered Care vs Measurement-Based Care; Three-way interaction effect (treatment, polynomial time, and SMI group). Participants with a diagnosis of major depression, schizoaffective or schizophrenia were classified into the SMI group and the reference group (Non-SMI) included diagnosis of anxiety, PTSD, depression/dysthymia/depression nos; Test type: Superiority; p = 0.3164, Mixed Models Analysis
Statistical Analysis 4: Comparison: Person-Centered Care vs Measurement-Based Care; Three-way interaction effect of time, treatment, and the basis subgroups (no symptoms =group 1; at least 1 severe symptom = group 2); Test type: Superiority; p = 0.0482, Mixed Models Analysis
Statistical Analysis 5: Comparison: Person-Centered Care vs Measurement-Based Care; Three-way interaction of Treatment, time, and subgroup of side effects. Subgroup of side effect= 0 if the response to the medication side effects question at baseline is 1, 2, or 3 (i.e. subgroup of participants who are minimally bothered by medication side effects at baseline); Subgroup of side effect= 1 if the response to the medication side effects question at baseline is 4-10 (i.e. subgroup of participants who are moderately or very bothered by medication side effects at baseline); Test type: Superiority; p = 0.9928, Mixed Models Analysis

2. Primary Outcome: Shared Decision Making Questionnaire (SDM-Q-9)
Description: The SDM-Q-9 is a 9-item self-report measure of the degree of shared decision making in clinical encounters. There are 6 possible responses ranging from: Completely Disagree (0) to Completely Agree (5). Raw score ranges from 0 to 45. Multiplication of the raw score by 20/9 provides a score forced (transformed) to range from 0 to 100, where 0 indicates the lowest possible level of SDM and 100 indicates the highest extent of shared decision making in clinical encounters. SDM-Q-9 scores for each time point reflect the mean score of all measures collected within that time frame.
Time Frame: Baseline and every eight months during the two-year intervention phase
Population: Multiple records can be measured from the same participant at the same time period, so N can be greater than the unique number of participants except for the baseline
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: Survey Records
Arm/Group | Person-Centered Care | Measurement-Based Care
Number analyzed (Participants) | 1201 | 1162
Number analyzed (Survey Records) | 3768 | 3705
Units on a scale
  Baseline: number analyzed (Participants) | 1197 | 1154
  Baseline: number analyzed (Survey Records) | 1197 | 1154
  Baseline | 74.082 (24.162) | 73.69 (24.271)
  Month 3: Every record 0< month <=3: number analyzed (Participants) | 5 | 3
  Month 3: Every record 0< month <=3: number analyzed (Survey Records) | 5 | 3
  Month 3: Every record 0< month <=3 | 72 (18.699) | 83.703 (8.411)
  Month 6: Every record 3< month <=6: number analyzed (Participants) | 222 | 189
  Month 6: Every record 3< month <=6: number analyzed (Survey Records) | 222 | 189
  Month 6: Every record 3< month <=6 | 75.946 (22.206) | 76.12 (21.756)
  Month 8: Every record 6< month <=8: number analyzed (Participants) | 301 | 245
  Month 8: Every record 6< month <=8: number analyzed (Survey Records) | 301 | 245
  Month 8: Every record 6< month <=8 | 74.692 (22.911) | 74.014 (22.852)
  Month 12: Every record 8< month <=12: number analyzed (Participants) | 265 | 296
  Month 12: Every record 8< month <=12: number analyzed (Survey Records) | 285 | 314
  Month 12: Every record 8< month <=12 | 76.148 (23.389) | 77.629 (19.988)
  Month16: Every record 12< month <=16: number analyzed (Participants) | 540 | 447
  Month16: Every record 12< month <=16: number analyzed (Survey Records) | 765 | 523
  Month16: Every record 12< month <=16 | 75.736 (21.823) | 76.325 (22.733)
  Month 18: Every record 16< month <=18: number analyzed (Participants) | 195 | 365
  Month 18: Every record 16< month <=18: number analyzed (Survey Records) | 204 | 405
  Month 18: Every record 16< month <=18 | 78.682 (21.648) | 76.554 (21.015)
  Month 20: Every record 18< month <=20: number analyzed (Participants) | 331 | 350
  Month 20: Every record 18< month <=20: number analyzed (Survey Records) | 383 | 380
  Month 20: Every record 18< month <=20 | 76.728 (19.737) | 75.72 (21.73)
  Month 24: Every record 20< month: number analyzed (Participants) | 337 | 417
  Month 24: Every record 20< month: number analyzed (Survey Records) | 406 | 492
  Month 24: Every record 20< month | 77.822 (20.898) | 77.082 (21.801)
Statistical Analysis 1: Comparison: Person-Centered Care vs Measurement-Based Care; Time-by-treatment interaction; Test type: Superiority; p = 0.6243, Mixed Models Analysis
Statistical Analysis 2: Comparison: Person-Centered Care vs Measurement-Based Care; Test for change over time from baseline (Marginal Effect of Time); Test type: Superiority; p = 0.1969, Mixed Models Analysis
Statistical Analysis 3: Comparison: Person-Centered Care vs Measurement-Based Care; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.0042, Mixed Models Analysis
Statistical Analysis 4: Comparison: Person-Centered Care vs Measurement-Based Care; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.0002, Mixed Models Analysis
Statistical Analysis 5: Comparison: Person-Centered Care vs Measurement-Based Care; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.7254, Mixed Models Analysis
Statistical Analysis 6: Comparison: Person-Centered Care vs Measurement-Based Care; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = 0.0580, Mixed Models Analysis

3. Secondary Outcome: Hope
Description: Patient hopefulness will be assessed using a single question: "Overall, how hopeful does the patient feel about his/her life?" Responses are on a scale of 1 through 10 with 1=No Hope and 10=Filled with Hope. Hopefulness scores for each time point reflect the mean score of all measures collected within that time frame.
Time Frame: Baseline and every eight months during the two-year intervention phase
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: Survey Records
Arm/Group | Person-Centered Care | Measurement-Based Care
Number analyzed (Participants) | 1201 | 1162
Number analyzed (Survey Records) | 3769 | 3706
Units on a scale
  Baseline: number analyzed (Participants) | 1196 | 1154
  Baseline: number analyzed (Survey Records) | 1196 | 1154
  Baseline | 6.008 (2.469) | 6.003 (2.413)
  Month 3: Every record 0< month <=3: number analyzed (Participants) | 4 | 3
  Month 3: Every record 0< month <=3: number analyzed (Survey Records) | 4 | 3
  Month 3: Every record 0< month <=3 | 6.5 (2.082) | 4 (1.732)
  Month 6: Every record 3< month <=6: number analyzed (Participants) | 219 | 189
  Month 6: Every record 3< month <=6: number analyzed (Survey Records) | 219 | 189
  Month 6: Every record 3< month <=6 | 6.078 (2.483) | 5.984 (2.303)
  Month 8: Every record 6< month <=8: number analyzed (Participants) | 301 | 246
  Month 8: Every record 6< month <=8: number analyzed (Survey Records) | 301 | 246
  Month 8: Every record 6< month <=8 | 6.073 (2.471) | 5.959 (2.439)
  Month 12: Every record 8< month <=12: number analyzed (Participants) | 268 | 295
  Month 12: Every record 8< month <=12: number analyzed (Survey Records) | 288 | 313
  Month 12: Every record 8< month <=12 | 6.118 (2.409) | 6.105 (2.338)
  Month16: Every record 12< month <=16: number analyzed (Participants) | 541 | 447
  Month16: Every record 12< month <=16: number analyzed (Survey Records) | 766 | 524
  Month16: Every record 12< month <=16 | 6.166 (2.413) | 6.164 (2.145)
  Month 18: Every record 16< month <=18: number analyzed (Participants) | 195 | 365
  Month 18: Every record 16< month <=18: number analyzed (Survey Records) | 204 | 405
  Month 18: Every record 16< month <=18 | 6.583 (2.176) | 6.185 (2.2)
  Month 20: Every record 18< month <=20: number analyzed (Participants) | 330 | 351
  Month 20: Every record 18< month <=20: number analyzed (Survey Records) | 382 | 381
  Month 20: Every record 18< month <=20 | 6.225 (2.245) | 6.092 (2.316)
  Month 24: Every record 20< month: number analyzed (Participants) | 340 | 416
  Month 24: Every record 20< month: number analyzed (Survey Records) | 409 | 491
  Month 24: Every record 20< month | 6.374 (2.348) | 6.312 (2.196)
Statistical Analysis 1: Comparison: Person-Centered Care vs Measurement-Based Care; Time-by-treatment interaction; Test type: Superiority; p = 0.4677, Mixed Models Analysis
Statistical Analysis 2: Comparison: Person-Centered Care vs Measurement-Based Care; Test for change over time from baseline (Marginal Effect of Time); Test type: Superiority; p = 0.0940, Mixed Models Analysis

4. Secondary Outcome: Medication Side Effects
Description: Medication side effects will be assessed using a single question: "How much is the patient troubled by medication side effects?" Responses are on a scale of 1 through 10 with 1=Not Bothered at all by side effects and 10=Very Bothered by side effects. Medication side effect scores for each time point reflect the mean score of all measures collected within that time frame.
Time Frame: Baseline and every eight months during the two-year intervention phase
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: Survey Records
Arm/Group | Person-Centered Care | Measurement-Based Care
Number analyzed (Participants) | 1201 | 1162
Number analyzed (Survey Records) | 3766 | 3702
Units on a scale
  Baseline: number analyzed (Participants) | 1194 | 1149
  Baseline: number analyzed (Survey Records) | 1194 | 1149
  Baseline | 3.935 (2.759) | 3.849 (2.746)
  Month 3: Every record 0< month <=3: number analyzed (Participants) | 4 | 3
  Month 3: Every record 0< month <=3: number analyzed (Survey Records) | 4 | 3
  Month 3: Every record 0< month <=3 | 3.75 (2.217) | 4.333 (3.215)
  Month 6: Every record 3< month <=6: number analyzed (Participants) | 220 | 189
  Month 6: Every record 3< month <=6: number analyzed (Survey Records) | 220 | 189
  Month 6: Every record 3< month <=6 | 3.527 (2.469) | 3.878 (2.654)
  Month 8: Every record 6< month <=8: number analyzed (Participants) | 302 | 246
  Month 8: Every record 6< month <=8: number analyzed (Survey Records) | 302 | 246
  Month 8: Every record 6< month <=8 | 3.884 (2.726) | 3.858 (2.82)
  Month 12: Every record 8< month <=12: number analyzed (Participants) | 268 | 295
  Month 12: Every record 8< month <=12: number analyzed (Survey Records) | 288 | 313
  Month 12: Every record 8< month <=12 | 3.67 (2.763) | 3.687 (2.738)
  Month16: Every record 12< month <=16: number analyzed (Participants) | 540 | 446
  Month16: Every record 12< month <=16: number analyzed (Survey Records) | 764 | 523
  Month16: Every record 12< month <=16 | 3.728 (2.67) | 3.717 (2.609)
  Month 18: Every record 16< month <=18: number analyzed (Participants) | 195 | 366
  Month 18: Every record 16< month <=18: number analyzed (Survey Records) | 204 | 406
  Month 18: Every record 16< month <=18 | 3.373 (2.674) | 3.502 (2.604)
  Month 20: Every record 18< month <=20: number analyzed (Participants) | 329 | 352
  Month 20: Every record 18< month <=20: number analyzed (Survey Records) | 381 | 382
  Month 20: Every record 18< month <=20 | 3.751 (2.745) | 3.72 (2.749)
  Month 24: Every record 20< month: number analyzed (Participants) | 340 | 417
  Month 24: Every record 20< month: number analyzed (Survey Records) | 409 | 491
  Month 24: Every record 20< month | 3.531 (2.705) | 3.595 (2.602)
Statistical Analysis 1: Comparison: Person-Centered Care vs Measurement-Based Care; Time-by-treatment interaction; Test type: Superiority; p = 0.8733, Mixed Models Analysis
Statistical Analysis 2: Comparison: Person-Centered Care vs Measurement-Based Care; Test for change over time from baseline (Marginal Effect of Time); Test type: Superiority; p = 0.0113, Mixed Models Analysis

5. Secondary Outcome: Patient Activation Measure (PAM)
Description: PAM is a 13-item scale that assesses the knowledge, skills, and confidence of patients essential to managing their own health and health care. Response options are: Strongly Disagree, Disagree, Agree, and Strongly Agree. The activation scale for the PAM ranges from 0 to 100. The lower values represent a poor outcome while higher values represent a better outcome. Overall possible range was 0 to 91.6. PAM scores for each time point reflect the mean score of all measures collected within that time frame.
Time Frame: Baseline and every eight months during the two-year intervention phase
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: Survey Records
Arm/Group | Person-Centered Care | Measurement-Based Care
Number analyzed (Participants) | 1201 | 1162
Number analyzed (Survey Records) | 3065 | 3081
Units on a scale
  Baseline: number analyzed (Participants) | 1006 | 987
  Baseline: number analyzed (Survey Records) | 1006 | 987
  Baseline | 62.707 (15.321) | 62.467 (15.635)
  Month 3: Every record 0< month <=3: number analyzed (Participants) | 4 | 3
  Month 3: Every record 0< month <=3: number analyzed (Survey Records) | 4 | 3
  Month 3: Every record 0< month <=3 | 47.75 (7.932) | 60.467 (7.81)
  Month 6: Every record 3< month <=6: number analyzed (Participants) | 187 | 153
  Month 6: Every record 3< month <=6: number analyzed (Survey Records) | 187 | 153
  Month 6: Every record 3< month <=6 | 63.979 (15.814) | 60.908 (14.959)
  Month 8: Every record 6< month <=8: number analyzed (Participants) | 260 | 195
  Month 8: Every record 6< month <=8: number analyzed (Survey Records) | 260 | 195
  Month 8: Every record 6< month <=8 | 62.978 (14.82) | 62.826 (15.275)
  Month 12: Every record 8< month <=12: number analyzed (Participants) | 210 | 245
  Month 12: Every record 8< month <=12: number analyzed (Survey Records) | 220 | 258
  Month 12: Every record 8< month <=12 | 63.205 (14.945) | 64.04 (16.678)
  Month16: Every record 12< month <=16: number analyzed (Participants) | 447 | 375
  Month16: Every record 12< month <=16: number analyzed (Survey Records) | 621 | 431
  Month16: Every record 12< month <=16 | 63.741 (14.852) | 63.034 (15.478)
  Month 18: Every record 16< month <=18: number analyzed (Participants) | 145 | 298
  Month 18: Every record 16< month <=18: number analyzed (Survey Records) | 152 | 328
  Month 18: Every record 16< month <=18 | 64.73 (14.668) | 63.413 (14.389)
  Month 20: Every record 18< month <=20: number analyzed (Participants) | 265 | 296
  Month 20: Every record 18< month <=20: number analyzed (Survey Records) | 304 | 319
  Month 20: Every record 18< month <=20 | 63.664 (14.593) | 63.642 (15.07)
  Month 24: Every record 20< month: number analyzed (Participants) | 264 | 351
  Month 24: Every record 20< month: number analyzed (Survey Records) | 311 | 407
  Month 24: Every record 20< month | 63.952 (14.887) | 63.895 (15.289)
Statistical Analysis 1: Comparison: Person-Centered Care vs Measurement-Based Care; Time-by-treatment interaction; Test type: Superiority; p = 0.2328, Mixed Models Analysis
Statistical Analysis 2: Comparison: Person-Centered Care; Test for change over time from baseline (Marginal Effect of Time); Test type: Superiority; p = 0.0005, Mixed Models Analysis

6. Secondary Outcome: Behavior and Symptom Identification Scale (BASIS-24)
Description: The BASIS-24 identifies a wide range of symptoms and problems that occur across the psychiatric diagnostic spectrum. There are 5 ordered responses either ranging from No Difficulty to Extreme Difficulty or from None of the Time to All of the Time. Each of 24 questions is scored on a 5 point scale (from 0 to 4 where 0 is the lowest severity and 4 is the highest). The overall BASIS-24 score is a weighted sum that is computed by multiplying the rating for each question by its weight and totaling the weighted ratings for each question. Overall possible range was 0 to 3.99. BASIS-24 scores for each time point reflect the mean score of all measures collected within that time frame.
Time Frame: Baseline and every eight months during the two-year intervention phase
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: Survey Records
Arm/Group | Person-Centered Care | Measurement-Based Care
Number analyzed (Participants) | 1201 | 1162
Number analyzed (Survey Records) | 3566 | 3527
Units on a scale
  Baseline: number analyzed (Participants) | 1126 | 1092
  Baseline: number analyzed (Survey Records) | 1126 | 1092
  Baseline | 1.496 (0.737) | 1.483 (0.726)
  Month 3: Every record 0< month <=3: number analyzed (Participants) | 4 | 2
  Month 3: Every record 0< month <=3: number analyzed (Survey Records) | 4 | 2
  Month 3: Every record 0< month <=3 | 1.418 (0.552) | 2.03 (0.622)
  Month 6: Every record 3< month <=6: number analyzed (Participants) | 210 | 181
  Month 6: Every record 3< month <=6: number analyzed (Survey Records) | 210 | 181
  Month 6: Every record 3< month <=6 | 1.291 (0.776) | 1.449 (0.666)
  Month 8: Every record 6< month <=8: number analyzed (Participants) | 277 | 237
  Month 8: Every record 6< month <=8: number analyzed (Survey Records) | 277 | 237
  Month 8: Every record 6< month <=8 | 1.386 (0.724) | 1.431 (0.767)
  Month 12: Every record 8< month <=12: number analyzed (Participants) | 256 | 280
  Month 12: Every record 8< month <=12: number analyzed (Survey Records) | 275 | 297
  Month 12: Every record 8< month <=12 | 1.324 (0.782) | 1.432 (0.739)
  Month16: Every record 12< month <=16: number analyzed (Participants) | 519 | 430
  Month16: Every record 12< month <=16: number analyzed (Survey Records) | 724 | 504
  Month16: Every record 12< month <=16 | 1.3 (0.724) | 1.362 (0.722)
  Month 18: Every record 16< month <=18: number analyzed (Participants) | 187 | 346
  Month 18: Every record 16< month <=18: number analyzed (Survey Records) | 194 | 386
  Month 18: Every record 16< month <=18 | 1.179 (0.696) | 1.357 (0.737)
  Month 20: Every record 18< month <=20: number analyzed (Participants) | 322 | 336
  Month 20: Every record 18< month <=20: number analyzed (Survey Records) | 372 | 363
  Month 20: Every record 18< month <=20 | 1.252 (0.709) | 1.299 (0.704)
  Month 24: Every record 20< month: number analyzed (Participants) | 322 | 396
  Month 24: Every record 20< month: number analyzed (Survey Records) | 384 | 465
  Month 24: Every record 20< month | 1.245 (0.699) | 1.305 (0.72)
Statistical Analysis 1: Comparison: Person-Centered Care vs Measurement-Based Care; Time-by-treatment interaction; Test type: Superiority; p = 0.0033, Mixed Models Analysis

7. Secondary Outcome: Sheehan Disability Scale
Description: The Sheehan Disability Scale measures the extent to which three major sectors in the person's life are impaired by psychiatric symptoms (work/school, social/leisure life, and family/home life). The 3 items are summed together to form a single measure of global functional impairment that ranges from 0 (unimpaired) to 30 (highly impaired). Sheehan Disability Scale scores for each time point reflect the mean score of all measures collected within that time frame.
Time Frame: Baseline and every eight months during the two-year intervention phase
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: Survey Records
Arm/Group | Person-Centered Care | Measurement-Based Care
Number analyzed (Participants) | 1201 | 1162
Number analyzed (Survey Records) | 3691 | 3590
Units on a scale
  Baseline: number analyzed (Participants) | 1148 | 1107
  Baseline: number analyzed (Survey Records) | 1148 | 1107
  Baseline | 10.514 (8.727) | 10.826 (8.761)
  Month 3: Every record 0< month <=3: number analyzed (Participants) | 4 | 3
  Month 3: Every record 0< month <=3: number analyzed (Survey Records) | 4 | 3
  Month 3: Every record 0< month <=3 | 13.5 (8.347) | 19 (8.185)
  Month 6: Every record 3< month <=6: number analyzed (Participants) | 222 | 190
  Month 6: Every record 3< month <=6: number analyzed (Survey Records) | 222 | 190
  Month 6: Every record 3< month <=6 | 9.536 (8.776) | 10.737 (8.585)
  Month 8: Every record 6< month <=8: number analyzed (Participants) | 301 | 244
  Month 8: Every record 6< month <=8: number analyzed (Survey Records) | 301 | 244
  Month 8: Every record 6< month <=8 | 10.385 (8.388) | 11.467 (9.167)
  Month 12: Every record 8< month <=12: number analyzed (Participants) | 264 | 284
  Month 12: Every record 8< month <=12: number analyzed (Survey Records) | 281 | 299
  Month 12: Every record 8< month <=12 | 9.142 (8.49) | 11.278 (9.057)
  Month16: Every record 12< month <=16: number analyzed (Participants) | 533 | 439
  Month16: Every record 12< month <=16: number analyzed (Survey Records) | 752 | 514
  Month16: Every record 12< month <=16 | 9.116 (8.005) | 10.226 (8.537)
  Month 18: Every record 16< month <=18: number analyzed (Participants) | 193 | 352
  Month 18: Every record 16< month <=18: number analyzed (Survey Records) | 201 | 390
  Month 18: Every record 16< month <=18 | 8.209 (7.957) | 10.154 (8.59)
  Month 20: Every record 18< month <=20: number analyzed (Participants) | 326 | 337
  Month 20: Every record 18< month <=20: number analyzed (Survey Records) | 377 | 367
  Month 20: Every record 18< month <=20 | 9.151 (8.175) | 9.662 (7.858)
  Month 24: Every record 20< month: number analyzed (Participants) | 339 | 402
  Month 24: Every record 20< month: number analyzed (Survey Records) | 405 | 476
  Month 24: Every record 20< month | 8.837 (7.767) | 9.716 (8.062)
Statistical Analysis 1: Comparison: Person-Centered Care vs Measurement-Based Care; Time-by-treatment interaction; Test type: Superiority; p = 0.1649, Mixed Models Analysis
Statistical Analysis 2: Comparison: Person-Centered Care vs Measurement-Based Care; Test for change over time from baseline (Marginal Effect of Time); Test type: Superiority; p = 0.0016, Mixed Models Analysis

8. Secondary Outcome: Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (QLESQ-SF)
Description: Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form is a 16-item, self-report questionnaire for assessing quality of life in multiple domains (e.g., physical health, mood, leisure time activities, social relationships, and overall). Response items are on a 5-point scale ranging from Very Poor to Very Good. The scoring of the Q-LES-Q-SF involves summing only the first 14 items to yield a raw total score. The last two items are not included in the total score but are standalone items. The raw total score ranges from 14 to 70. The raw total score was transformed into a percentage maximum possible score using the following formula. The lower values/percentages represent a poor outcome while higher values/percentages represent a better outcome. Overall possible range was 0-100. QLESQ-SF scores for each time point reflect the mean score of all measures collected within that time frame.
Time Frame: Baseline and every eight months during the two-year intervention phase
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: Survey Records
Arm/Group | Person-Centered Care | Measurement-Based Care
Number analyzed (Participants) | 1201 | 1162
Number analyzed (Survey Records) | 3398 | 3359
Units on a scale
  Baseline: number analyzed (Participants) | 1039 | 1024
  Baseline: number analyzed (Survey Records) | 1039 | 1024
  Baseline | 54.922 (21.316) | 53.51 (20.758)
  Month 3: Every record 0< month <=3: number analyzed (Participants) | 3 | 3
  Month 3: Every record 0< month <=3: number analyzed (Survey Records) | 3 | 3
  Month 3: Every record 0< month <=3 | 52.38 (16.003) | 37.5 (14.616)
  Month 6: Every record 3< month <=6: number analyzed (Participants) | 201 | 176
  Month 6: Every record 3< month <=6: number analyzed (Survey Records) | 201 | 176
  Month 6: Every record 3< month <=6 | 57.756 (21.417) | 52.902 (21.231)
  Month 8: Every record 6< month <=8: number analyzed (Participants) | 280 | 232
  Month 8: Every record 6< month <=8: number analyzed (Survey Records) | 280 | 232
  Month 8: Every record 6< month <=8 | 57.417 (20.472) | 53.271 (22.152)
  Month 12: Every record 8< month <=12: number analyzed (Participants) | 247 | 272
  Month 12: Every record 8< month <=12: number analyzed (Survey Records) | 264 | 286
  Month 12: Every record 8< month <=12 | 59.037 (21.651) | 54.383 (20.661)
  Month16: Every record 12< month <=16: number analyzed (Participants) | 495 | 403
  Month16: Every record 12< month <=16: number analyzed (Survey Records) | 694 | 471
  Month16: Every record 12< month <=16 | 58.018 (20.553) | 54.375 (20.337)
  Month 18: Every record 16< month <=18: number analyzed (Participants) | 176 | 328
  Month 18: Every record 16< month <=18: number analyzed (Survey Records) | 183 | 365
  Month 18: Every record 16< month <=18 | 62.754 (20.621) | 54.31 (19.872)
  Month 20: Every record 18< month <=20: number analyzed (Participants) | 312 | 319
  Month 20: Every record 18< month <=20: number analyzed (Survey Records) | 359 | 345
  Month 20: Every record 18< month <=20 | 60.396 (20.464) | 55.192 (20.609)
  Month 24: Every record 20< month: number analyzed (Participants) | 317 | 385
  Month 24: Every record 20< month: number analyzed (Survey Records) | 375 | 457
  Month 24: Every record 20< month | 59.881 (20.056) | 56.666 (20.068)
Statistical Analysis 1: Comparison: Person-Centered Care vs Measurement-Based Care; Time-by-treatment interaction; Test type: Superiority; p = 0.0080, Mixed Models Analysis

9. Secondary Outcome: Engagement in Medication and Evaluation Visit
Description: Count of the number of medication checks and evaluation visits for each study participant for the 12 month period prior to and including the anchor date of the time point.
Time Frame: Baseline, 8 months, 24 months
Population: Based on participants who had available claims data.
Measure: Mean (Standard Deviation); unit: medication checks and evaluation visits
Arm/Group | Person-Centered Care | Measurement-Based Care
Number analyzed (Participants) | 1064 | 1045
medication checks and evaluation visits
  Baseline: number analyzed (Participants) | 1064 | 1000
  Baseline | 6.356 (4.22) | 6.785 (4.006)
  8 months: number analyzed (Participants) | 1059 | 1045
  8 months | 5.977 (4.586) | 6.851 (3.94)
  24 months: number analyzed (Participants) | 996 | 976
  24 months | 5.517 (4.803) | 5.691 (4.839)
Statistical Analysis 1: Comparison: Person-Centered Care vs Measurement-Based Care; Test type: Superiority; p < 0.0001, Mixed Models Analysis

10. Secondary Outcome: Engagement in Psychotherapy Visit
Description: Count of the number of psychotherapy visits for each study participant for the 12 month period prior to and including the anchor date of the time point.
Time Frame: Baseline, 8 months, 24 months
Population: Based on participants who had available claims data.
Measure: Mean (Standard Deviation); unit: psychotherapy visits
Arm/Group | Person-Centered Care | Measurement-Based Care
Number analyzed (Participants) | 1064 | 1045
psychotherapy visits
  Baseline: number analyzed (Participants) | 1064 | 1000
  Baseline | 8.706 (12.972) | 9.679 (12.313)
  8 months: number analyzed (Participants) | 1059 | 1045
  8 months | 7.825 (12.461) | 9.369 (12.279)
  24 months: number analyzed (Participants) | 996 | 976
  24 months | 7.224 (12.728) | 6.864 (11.397)
Statistical Analysis 1: Comparison: Person-Centered Care vs Measurement-Based Care; Test type: Superiority; p = 0.0003, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Over the 24-month intervention period.
Description: This is a behavioral intervention that did not involve "Serious" and "Other" adverse events, hence the reason none are reported.
Groups:
- Person-Centered Care: Decision support center staffed by peers. Patient uses the CommonGround program prior to medication visit to prepare a personal report, with support from peer(s). The CommonGround report expresses goals for medication, how other strategies help with functioning, current problems, and medication side effects. Patient brings report into the medication visit. Prescriber and patient discuss medication options, and prescriber enters the shared decision into CommonGround during the visit. Person-Centered Care: Decision support center staffed by peers. Patient uses the CommonGround program prior to medication visit to prepare a personal report, with support from peer(s). The CommonGround report expresses goals for medication, how other strategies help with functioning, current problems, and medication side effects. Patient brings report into the medication visit. Prescriber and patient discuss medication options, and prescriber enters the shared decision into CommonGround during the visit.
Arm/Group | Person-Centered Care | Measurement-Based Care
All-Cause Mortality (participants affected / at risk) | 12/1232 | 16/1211
Serious Adverse Events (participants affected / at risk) | 0/1232 | 0/1211
Other Adverse Events (participants affected / at risk) | 0/1232 | 0/1211

LIMITATIONS AND CAVEATS:
The PEMM was developed for this study. For unavoidable reasons, site randomization was not maintained. Data collection timepoints were expanded.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No